CLINICAL TRIAL: NCT00548340
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Investigate the Efficacy and Safety of VEC-162 (20 mg/Day and 50 mg/Day) in the Treatment of Primary Insomnia
Brief Title: VEC-162 Study in Adult Patients With Primary Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-VEC-162-3104
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- VEC-162 20 mg (Experimental): VEC-162 (tasimelteon) 20 mg capsules PO daily for five weeks
  Interventions: Drug: VEC-162 20 mg
- VEC-162 50 mg (Experimental): VEC-162 (tasimelteon) 50 mg capsules PO daily for five weeks
  Interventions: Drug: VEC-162 50 mg
- Placebo (Placebo Comparator): Placebo capsules PO daily five weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VEC-162 20 mg — 20 mg VEC-162 (tasimelteon) capsules, PO daily for five weeks
  Arms: VEC-162 20 mg
Drug: Placebo — Placebo capsules, PO daily for five weeks
  Arms: Placebo
Drug: VEC-162 50 mg — 50 mg VEC-162 (tasimelteon) capsules, PO daily for five weeks
  Arms: VEC-162 50 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a 5 week double-blind treatment period of VEC-162 as compared to placebo in male and female patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with a diagnosis of primary insomnia as defined in DSM-IV.
* Habitual bedtime between 9:00 pm and 1:00 am.
* No history or evidence of restless leg syndrome or periodic limb movement disorder or sleep apnea.
* Patients must sign a written consent form.

Exclusion Criteria:

* History of drug or alcohol abuse as defined in DSM-IV.
* History of psychiatric disorders, including Major Depressive Disorder, Generalized Anxiety Disorder and delirium.
* History of chronic obstructive pulmonary disease (COPD), seizures, sleep apnea, narcolepsy, circadian-rhythm sleep disorder, parasomnia or any sleep disorder other than chronic insomnia.
* Recent history of shift work or jet lag.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 322 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Vanda Investigational Site, Birmingham, Alabama
  - Vanda Investigational Site, Hot Springs, Arkansas
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Anaheim, California
  - Vanda Investigational Site, Burbank, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Colorado Springs, Colorado
  - Vanda Investigational Site, Hallandale, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Naples, Florida
  - Vanda Investigational Site, Orlando, Florida
  - Vanda Investigational Site, Pembroke Pines, Florida
  - Vanda Investigational Site, St. Petersburg, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Chicago, Illinois
  - Vanda Investigational Site, Overland Park, Kansas
  - Vanda Investigational Site, Crestview Hills, Kentucky
  - Vanda Investigational Site, Lexington, Kentucky
  - Vanda Investigational Site, Louisville, Kentucky
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, Newton, Massachusetts
  - Vanda Investigational Site, Troy, Michigan
  - Vanda Investigational Site, Chesterfield, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, West Seneca, New York
  - Vanda Investigational Site, Raleigh, North Carolina
  - Vanda Investigational Site, Beachwood, Ohio
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Oklahoma City, Oklahoma
  - Vanda Investigational Site, Columbia, South Carolina
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- VEC-162 20 mg: VEC-162: 20 mg VEC-162 capsules, PO daily for five weeks
- VEC-162 50 mg: VEC-162: 50 mg VEC-162 capsules, PO daily for five weeks
Period: Overall Study
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Started | 109 | 109 | 104
Completed | 101 | 98 | 95
Not Completed | 8 | 11 | 9
Not completed — Protocol Violation | 2 | 3 | 3
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 3
Not completed — Other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo | Total
Number analyzed (Participants) | 109 | 109 | 104 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.6) | 40.7 (10.4) | 41.7 (11.8) | 41.8 (10.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 109 | 104 | 322
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 63 | 68 | 197
  Male | 43 | 46 | 36 | 125

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline - Latency to Persistent Sleep (LPS)
Description: Average latency to persistent sleep is defined as the length of time elapsed between lights off and onset of persistent sleep (defined as the point at which 10 minutes of uninterrupted sleep has begun as determined by PSG) between Baseline and the average of nights 1 and 8.
Time Frame: Baseline, Night 1, and Night 8 measurement
Population: One subject randomized to VEC-162 20 mg did not have any post-baseline PSG data and was excluded from the Full Analysis Population.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Number analyzed (Participants) | 108 | 109 | 104
minutes | 45.0 (2.965) | 46.4 (2.954) | 28.3 (3.020)

2. Secondary Outcome: Average Change From Baseline - Wake After Sleep Onset (WASO) and Total Sleep Time (TST)
Description: Average wake after sleep onset was defined as the time spent awake between onset of sleep (latency to non-awake) and lights-on, as determined by PSG between Baseline, and the average of nights 1 and 8. Total sleep time (TST) was defined as the time spent sleeping between lights-out and lights-on, i.e., full night between Baseline, and the average of nights 1 and 8.
Time Frame: Baseline, Night 1, and Night 8 measurements for WASO and TST
Population: One subject randomized to VEC-162 20 mg did not have post-baseline PSG data and was excluded from the Full Analysis population.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Number analyzed (Participants) | 108 | 109 | 104
minutes
  Avg WASO Change from Baseline | 12.2 (4.349) | 14.1 (4.329) | 11.7 (4.569)
  Avg TST Change from Baseline | 51.4 (4.794) | 52.0 (4.775) | 39.9 (4.882)

3. Post Hoc Outcome: Average Change From Baseline - Latency to Persistent Sleep (LPS)
Description: Average latency to persistent sleep is defined as the length of time elapsed between lights off and onset of persistent sleep (defined as the point 10 minutes of uninterrupted sleep has begun as determined by PSG) between Baseline, and the average of nights 22 and 29.
Time Frame: Baseline, Night 22, and Night 29 measurement
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Number analyzed (Participants) | 108 | 109 | 104
minutes | 49.4 (3.309) | 45.1 (3.292) | 33.9 (3.338)

4. Post Hoc Outcome: Average Change From Baseline - Wake After Sleep Onset (WASO) and Total Sleep Time (TST)
Description: Average wake after sleep onset was defined as the time spent awake between onset of sleep (latency to non-awake) and lights-on, as determined by PSG between Baseline, and the average of nights 22 and 29. Total sleep time (TST) was defined as the time spent sleeping between lights-out and lights-on, i.e., full night between Baseline, and the average of nights 22 and 29.
Time Frame: Baseline, Night 22, and Night 29 measurements for WASO and TST
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Number analyzed (Participants) | 108 | 109 | 104
minutes
  Avg WASO Change from Baseline | 17.7 (4.139) | 10.2 (4.184) | 20.3 (4.381)
  Avg TST Change from Baseline | 60.3 (4.821) | 48.6 (4.802) | 47.4 (4.882)

ADVERSE EVENTS:
Time Frame: Night 1 to Day 37 (EOS)
Arm/Group | VEC-162 20 mg | VEC-162 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/109 | 0/109 | 1/104
Other Adverse Events (participants affected / at risk) | 15/109 | 13/109 | 11/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEC-162 20 mg (N=109) | VEC-162 50 mg (N=109) | Placebo (N=104)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEC-162 20 mg (N=109) | VEC-162 50 mg (N=109) | Placebo (N=109)
Headache (Nervous system disorders) | 11 (14) | 4 (4) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 5 (5) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No